CLINICAL TRIAL: NCT04970628
Title: Risk Factors Analysis and Evaluation System Construction of Airway Obstruction After Anterior Cervical Surgery
Brief Title: Risk Factors Analysis After Anterior Cervical Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020406
Record Dates: First submitted 2021-07-01; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cervical Spondylosis
Keywords: Cervical Spondylosis; Anterior cervical surgery; Postoperative airway obstruction
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients performed airway obstruction after anterior cervical operation
  Interventions: Other: Medical records collection
- Control group: Patients did not perform airway obstruction after anterior cervical operation
  Interventions: Other: Medical records collection

INTERVENTIONS:
Other: Medical records collection — Patient's medical records before and after surgery.

SUMMARY:
This study is to collect and summarize the cases of airway obstruction after anterior cervical operation through retrospective case analysis, to explore the risk factors of airway obstruction after anterior cervical operation, to provide the basis for the construction of evaluation system and provide reference for the nursing of postoperative complications.

DETAILED DESCRIPTION:
1. Research objects The clinical data of patients who underwent anterior cervical surgery in our department from 2010 to 2019 were retrospectively collected. The cases of patients who underwent reoperation and those who did not underwent reoperation and the causes of airway obstruction were analyzed. They were evaluated by ward doctors, anesthesiologists and ward nurses according to clinical standards. The following inclusion and exclusion criteria were used. Inclusion criteria: patients undergoing anterior cervical surgery from 2010 to 2019; Age ≥ 18 years old. Exclusion criteria: age ≤ 18 years old; Patients with neck tumor, infection and goiter; Neck soft tissue and bone structure deformity; Ankylosing spondylitis; Oral and laryngopharyngeal diseases; Hysteria or mental illness; Postoperative anesthesia can not be normal resuscitation patients; Nervous system diseases: such as Parkinson's disease. Patients with airway obstruction due to epidural hematoma underwent reoperation.

   Grouping of patients:①Case group: patients who underwent anterior cervical spine surgery from 2010 to 2019 and had airway obstruction and re intubation in a short time after surgery. ②Control group: among the patients who never had reoperation of postoperative airway obstruction, the number of cases closest to this time point was collected according to the maximum matching ratio of 1:4 according to the operation time of patients in case group.
2. Research methods The exposure history of various possible risk factors in the past was collected by inquiring and consulting medical records. Through literature review, the most direct cause of airway obstruction after anterior cervical surgery is the compression of trachea caused by neck hematoma, the increase of respiratory secretions, airway obstruction, dyspnea and even asphyxia. In the research of Li Haoxi, Chen Xiongsheng and other experts, it is pointed out that the age, smoking, body mass index, hypertension, operation mode, operation time and number of operation segments of patients have a significant impact on the airway obstruction after anterior cervical surgery, which is consistent with some foreign related reports. The risk of airway obstruction in smokers and those aged 60 or above increased significantly compared with those who did not smoke and <45 years old. Meanwhile, the incidence rate of chronic pharyngitis in smokers was significantly higher than that in non-smokers. With the increase of smoking time and age, chronic pharyngitis was also a high-risk factor. According to the statistical results of the study, the incidence of re intubation of airway obstruction after single segment anterior cervical surgery was 0.3%, and the incidence of airway obstruction was 4.97% with the increase of surgical segments. Studies suggest that prevention of hematoma, intraoperative clear exposure and thorough hemostasis are the first factors, and treatment of possible active bleeding. In the study, a case of hematoma in a patient with hypertension was taken as an example to point out that patients with hypertension will have the risk of bleeding again after operation. When the patient has obvious obesity, the neck is short and thick in appearance, and tissue edema is easy to occur after operation, resulting in drainage affected. ①preoperative assessment: age, gender, height, weight (BMI), smoking history, drinking history, hypertension, diabetes mellitus, chronic pharyngitis, neck circumference and sleep monitoring.

   * Intraoperative factors: operation mode, operation segment location, operation time, intraoperative blood loss, anesthesia recovery time. ③Postoperative evaluation: respiratory condition, blood oxygen, blood pressure, drainage volume, limb muscle strength, expectoration.

In order to explore the relationship between risk factors and airway obstruction, the exposure proportion of each index in case group and control group was compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing anterior cervical surgery from 2010 to 2019;
* Age ≥ 18 years old.

Exclusion Criteria:

* Age ≤ 18 years old;
* Patients with neck tumor, infection and goiter;
* Neck soft tissue and bone structure deformity;
* Ankylosing spondylitis;
* Oral and laryngopharyngeal diseases;
* Hysteria or mental illness;
* Postoperative anesthesia can not be normal resuscitation patients;
* Nervous system diseases: such as Parkinson's disease.
* Patients with airway obstruction due to epidural hematoma underwent reoperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical data of patients who underwent anterior cervical surgery in our department from 2010 to 2019 were retrospectively collected. The cases of patients who underwent reoperation and those who did not underwent reoperation and the causes of airway obstruction were analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic data | Before surgery
  Age, gender, height, weight (BMI), smoking history, drinking history, hypertension, diabetes mellitus
Data about operation | During surgery
  Operation method
Data about operation | During surgery
  Operative section location
Data about operation | During surgery
  Operation time
Data about operation | During surgery
  Blood loss during operation
Data about operation | During surgery
  Recovery time of anesthesia
Postoperative data | After surgery to discharge, an average of 1 day
  Postoperative blood pressure
Postoperative data | After surgery to discharge, an average of 1 day
  Drainage volume

SECONDARY OUTCOMES:
History and evaluation | Before surgery
  Chronic pharyngitis
History and evaluation | Before surgery
  Sleep monitoring
Postoperative management | After surgery to discharge, an average of 1 day
  Neck circumference
Postoperative management | After surgery to discharge, an average of 1 day
  Expectoration

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No